CLINICAL TRIAL: NCT05390034
Title: REFLEX: A Randomized Controlled Trial to Test the Efficacy of an Emotion Regulation Flexibility Program With Daily Measures
Brief Title: Improving Emotion Regulation Flexibility: Testing the Efficacy of an Emotion Regulation Program in College Students
Acronym: REFLEX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Collaborators: University Grenoble Alps (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-A00378-35
Record Dates: First submitted 2022-03-17; First posted 2022-05-25 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-03

CONDITIONS: Anxiety Depression; Emotion Regulation
Keywords: emotion regulation flexibility; randomized controlled trial; experience sampling method; daily measures; emotion regulation program
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Intervention Model Description: Treatment compared to an active control group (i.e., a relaxation program group)
Who Masked: Participant
Masking Description: Participants will be randomized to one of the two arms (i.e., ART program or active control group). Outcomes assessments will be performed with online questionnaires.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ART (Experimental): Developed by Berking and Whitley (Berking & Whitley, 2014), this transdiagnostic program aims to improve general emotion regulation skills, and more specifically by increasing participants' emotion regulation flexibility. ART targets several skills, such as acceptance, tolerance, non-judgmental awareness, self-support, analysis of the causes of emotions and emotional modification. This intervention consists of 9 sessions (2 hours each), each of which starts with the presentation of a vicious circle for psycho-education. This vicious circle is then transformed into a virtuous circle by introducing an emotion regulation skill. Participants are invited to reflect, discuss and practice this skill. Exercises are also recommended at home, with the help of audios and a written workbook made available. All the material was translated into French for the purpose of this research.
  Interventions: Behavioral: ART
- Relaxation (Active Comparator): The relaxation group will be based mainly on the intervention developed by Dominique Servant (Relaxation and meditation, 2021), adapted for this research for the group format and divided into 9 modules (2 hours each). This intervention proposes an added psycho-education part similar to the dedicated session of the ART program, followed by the teaching of different relaxation techniques to the participants, who are invited to test them in session and then to practice them at home. This control group focuses on a specific component present in the ART group (relaxation), allowing us to assess the impact of the other components of the ART program and thus explore our flexibility hypothesis (requiring several emotion regulation skills). Note that the mindfulness meditation components were removed from the program for this study, as they were considered a second emotion regulation skill.
  Interventions: Behavioral: Relaxation

INTERVENTIONS:
Behavioral: ART — Session 1: Description of the group & Psychoeducation Session 2: Breathing and muscle relaxation Session 3: Importance of practice/motivation Session 4: Nonjudgemental awareness Session 5: Acceptance and tolerance Session 6: Self-support Session 7: Analysis of emotions Session 8: Modification of emotions Session 9: Practice and contextual applications + end of group
  Arms: ART
Behavioral: Relaxation — Session 1: Description of the groupe & Psychoeducation Session 2: Breathing control 1 Session 3: Breathing control 2 Session 4: Muscle relaxation Session 5: Visualisation Session 6: Stretching Session 7: Schultz relaxation Session 8: Schultz relaxation Session 9: Summary and end of group
  Arms: Relaxation

SUMMARY:
The main objective of this RCT is to test the efficacy of an emotion regulation group program (i.e., ART program) in college students, compared to an active control group (i.e., relaxation program). Using multilevel analyses, we expect an improvement in anxious-depressive symptomatology for both groups. However, we expect the ART group to improve specifically on emotion regulation flexibility ability, and the last to be a mediative variable on mental health.

DETAILED DESCRIPTION:
Emotion regulation (ER) is a process associated with difficulties in mental health. Given its transdiagnostic features, its improvement could facilitate the recovery of various psychological issues. A limit of current studies is the lack of knowledge regarding whether available interventions improve ER flexibility (i.e., the ability to implement ER strategies in line with contextual demands), even though this capacity has been associated with better mental health and well-being. Therefore, the aim of the study is to test the efficacy of a 9-weeks ER group program (the Affect Regulation Training-ART), using the most appropriate measures (i.e., experience sampling method) in a student population. Plus, the goal of the study is to explore the potential mediative role of ER flexibility on mental health improvement.

This RCT will compare the ART program group to an active control group (a relaxation program) in 100 participants. To test the mediative role of ER flexibility on mental health, daily measures will be used before, during, and after the interventions to evaluate the extent to which participants are flexible in their ER.

Using multilevel analyses, we expect an improvement in anxious-depressive symptomatology for both groups. However, we expect the ART group to improve specifically on ER flexibility ability, and the last to be a mediative variable on mental health.

This study will enhance knowledge on interventions for students and the impact of interventions on ER flexibility. Also, this research will improve knowledge on ecological measures for assessing the effect of interventions. Overall, this project represents new opportunities to improve ER skills to improve mental health in undergraduate students.

ELIGIBILITY:
Inclusion Criteria:

* Grenoble Alpes University student
* Having a smartphone that can host PIEL application
* BDI ≥ 10 and ≤ 30
* Reading, understanding, and speaking French
* Signed free and informed consent

Non inclusion Criteria:

* Participation in another study related to emotion regulation
* Participation in other psychotherapies involving cognitive and behavioral intervention (actual or in the past year)
* Changes in drug treatments in the last two months
* Student in psychology
* Individuals concerned in the articles L1121-6 à L1121-8 of CSP (i.e., protected individuals)
* Suicidal risk (BDI II, item suicidal thoughts > 1 or MINI suicide, low intensity)
* Anorexia nervose (MINI)
* Schizophrenic spectrum disorder (MINI)
* Substance abuse (heroin, cocaine, ecstasy) (MINI)

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 94 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Emotion regulation | 30 minutes
  Emotion Regulation Skills Questionnaire (score), higher scores mean better outcome, value minimum of 0 maximum 108

SECONDARY OUTCOMES:
Change in Depressive symptoms | 20 minutes
  Beck Depressive Inventory Questionnaire (BDI-II) (score), higher scores mean worse outcome, value minimum of 0 maximum 63
Change in Anxious symptoms | 20 minutes
  Beck Anxiety Inventory Questionnaire (BAI) (score), higher scores mean worse outcome, value minimum of 0 maximum 63
Change in Daily Emotion regulation flexibility | Immediately after the intervention
  Experience sampling method using PIEL application (flexibility in emotion regulation strategies) - Questionnaire on smartphone (score aggregated with the 3 times of measurements)

OTHER OUTCOMES:
Therapeutic alliance | During the procedure/Immediately after the intervention
  California Psychotherapy Alliance Scale - Control in the two groups - value minimum 24, maximum 168, higher scores mean better outcome
Expectancies on treatment | During the procedure
  Credibility and Expectancy Questionnaire - Control in the two groups, value minimum 4, maximum 36, higher scores mean better outcome
Changes in treatment | During the procedure/Immediately after the intervention
  Question on possible changes in psychological or drug treatment during intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Université Grenoble Alpes, Grenoble, France

IPD SHARING:
Plan to Share IPD: Yes
Theoretical background, objectives, hypothesis, expected results, methodology
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: 3 years
URL: http://osf.io/28xh6/

REFERENCES:
- [Result] Berking M, Eichler E, Luhmann M, Diedrich A, Hiller W, Rief W. Affect regulation training reduces symptom severity in depression - A randomized controlled trial. PLoS One. 2019 Aug 29;14(8):e0220436. doi: 10.1371/journal.pone.0220436. eCollection 2019. PMID 31465443
- [Result] Aldao A, Nolen-Hoeksema S. The influence of context on the implementation of adaptive emotion regulation strategies. Behav Res Ther. 2012 Aug;50(7-8):493-501. doi: 10.1016/j.brat.2012.04.004. Epub 2012 May 7. PMID 22659159
- [Result] Aldao A, Nolen-Hoeksema S, Schweizer S. Emotion-regulation strategies across psychopathology: A meta-analytic review. Clin Psychol Rev. 2010 Mar;30(2):217-37. doi: 10.1016/j.cpr.2009.11.004. Epub 2009 Nov 20. PMID 20015584
- [Result] Csikszentmihalyi M, Larson R. Validity and reliability of the Experience-Sampling Method. J Nerv Ment Dis. 1987 Sep;175(9):526-36. doi: 10.1097/00005053-198709000-00004. PMID 3655778
- [Result] Gross JJ. Emotion regulation: affective, cognitive, and social consequences. Psychophysiology. 2002 May;39(3):281-91. doi: 10.1017/s0048577201393198. PMID 12212647
- [Result] Kazdin AE. Mediators and mechanisms of change in psychotherapy research. Annu Rev Clin Psychol. 2007;3:1-27. doi: 10.1146/annurev.clinpsy.3.022806.091432. PMID 17716046